CLINICAL TRIAL: NCT04992988
Title: Concurrent Chemoradiotherapy With Toripalimab for Local-regional Recurrent Nasopharyngeal Carcinoma: a Prospective, Single-arm, Phase II Trial
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cancer Hospital of Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Song Qu, Principal Investigator, Cancer Hospital of Guangxi Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2020163
Record Dates: First submitted 2021-07-18; First posted 2021-08-06 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Nasopharyngeal Carcinoma; Toripalimab; Recurrent Nasopharyngeal Squamous Cell Carcinoma
Keywords: Nasopharyngeal Carcinoma; Toripalimab
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toripalimab+CCRT (Experimental): Cisplatin 100mg/m2(every three weeks),D1,D22,D43 of intensity modulated radiotherapy.
  Toripalimab 240mg every 3 weeks with a total of 3 cycles as concurrent anti-PD-1 immunotherapy; Toripalimab240mg every 3 weeks with a total of 9 cycles as adjuvant anti-PD-1 immunotherapy 3 weeks after CCRT
  Interventions: Drug: Toripalimab

INTERVENTIONS:
Drug: Toripalimab — Toripalimab 240mg every 3 weeks with a total of 3 cycles as concurrent anti-PD-1 immunotherapy; Toripalimab240mg every 3 weeks with a total of 9 cycles as adjuvant anti-PD-1 immunotherapy 2 weeks after CCRT

SUMMARY:
This is a prospective, single-arm, phase II trial to study the efficacy of PD-1 antibody Toripalimab combined with concurrent cisplatin chemoradiotherapy in treating patients with locoregionally recurrent nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly histologically confirmed recurrent nasopharyngeal carcinoma, or Two or more image examinations (MRI, and PET-CT) show the recurrence tumor
2. staged as rT3-4N0-1M0或rT1-4N2-3M0 （according to the 8th AJCC edition）
3. Satisfactory performance status: ECOG (Eastern Cooperative OncologyGroup) scale 0-1
4. Neutrophil ≥ 1.5×109 /L and PLT ≥4×109 /L and HGB ≥90 g/L
5. With normal liver function test (ALT、AST ≤ 2.5×ULN, TBIL≤ 1.5×ULN)
6. With normal renal function test ( creatinine clearance ≥60 ml/min)
7. sign an "informed consent form
8. Male and no pregnant female

Exclusion Criteria:

1. Age> 70, or < 18 years old
2. Hepatitis B surface antigen (HBsAg) positive and HBV-DNA ≥200IU/ml, or 1000cps/ml.
3. Patients with positive HCV antibody.
4. Active, known or suspected autoimmune disease; Type I Diabetes, hypothyroidism those only need hormone replacement therapy, and skin disease (leukoderma, psoriasis, alopecia et al) who don't need systemic therapy can recruit.
5. History of interstitial lung disease
6. Equivalent dose more than prednisone 10mg/d or other immunosuppressive treatments within 28 days prior to signing the informed consent.
7. Receive or will receive live vaccine within 30 days prior to signing the informed consent.
8. Women of child-bearing potential who are pregnant or breastfeeding.
9. Suffered from malignant tumors, except the carcinoma in situ, papillary thyroid carcinoma, or skin cancer (non- melanoma) within five years.
10. Hypersensitivity to macromolecular protein, or to any component of triplezumab.
11. HIV positive.
12. Severe, uncontrolled medical conditions and infections.
13. Other diseases which may influence the safety or compliance of the clinical trial, such as heart failure with symptom, unstable angina, myocardial infarction, active infections those need systemic therapy, mental illness, or their family and society factors.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-06-28 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2 years
  Defined from date of randomization to date of first documentation of death from any cause or censored at the date of the last follow-up.

SECONDARY OUTCOMES:
Progress-free survival (PFS) | 2 years
  Defined from date of randomization to date of first documentation of progression or death due to any cause.
Objective Response Rate （ORR） | After the completion of the PD-1 antibody and chemoradiotherapy treatment
  An objective response is defined as either a confirmed CR or a PR, as determined by the investigator using RECIST v1.1Response Evaluation Criteria in Solid Tumors (RECIST) from the National Cancer Institute (NCI).
Incidence rate of adverse events (AEs) | 2 years
  Analysis of adverse events (AEs) are based on treatment-related AEs (trAEs) and immune-related AEs (irAEs), and all-grade AEs and grade 3-4 AEs. AEs are evaluated by investigators according to the Common Terminology Criteria for Adverse Events, version 5.0
Change of QoL (quality of life) | 1 year
  QoL scores were assessed by using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire C30 (EORTCQLQ-C30) before radiotherapy, at the end of radiotherapy, at 12 months after radiotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangxi Medical University Cancer Hospital, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chen BJ, Chapuy B, Ouyang J, Sun HH, Roemer MG, Xu ML, Yu H, Fletcher CD, Freeman GJ, Shipp MA, Rodig SJ. PD-L1 expression is characteristic of a subset of aggressive B-cell lymphomas and virus-associated malignancies. Clin Cancer Res. 2013 Jul 1;19(13):3462-73. doi: 10.1158/1078-0432.CCR-13-0855. Epub 2013 May 14. PMID 23674495
- [Background] Fang W, Zhang J, Hong S, Zhan J, Chen N, Qin T, Tang Y, Zhang Y, Kang S, Zhou T, Wu X, Liang W, Hu Z, Ma Y, Zhao Y, Tian Y, Yang Y, Xue C, Yan Y, Hou X, Huang P, Huang Y, Zhao H, Zhang L. EBV-driven LMP1 and IFN-gamma up-regulate PD-L1 in nasopharyngeal carcinoma: Implications for oncotargeted therapy. Oncotarget. 2014 Dec 15;5(23):12189-202. doi: 10.18632/oncotarget.2608. PMID 25361008
- [Background] Dong H, Chen L. B7-H1 pathway and its role in the evasion of tumor immunity. J Mol Med (Berl). 2003 May;81(5):281-7. doi: 10.1007/s00109-003-0430-2. Epub 2003 Apr 30. PMID 12721664
- [Background] Pardoll DM. The blockade of immune checkpoints in cancer immunotherapy. Nat Rev Cancer. 2012 Mar 22;12(4):252-64. doi: 10.1038/nrc3239. PMID 22437870
- [Background] Ferris RL, Blumenschein G Jr, Fayette J, Guigay J, Colevas AD, Licitra L, Harrington K, Kasper S, Vokes EE, Even C, Worden F, Saba NF, Iglesias Docampo LC, Haddad R, Rordorf T, Kiyota N, Tahara M, Monga M, Lynch M, Geese WJ, Kopit J, Shaw JW, Gillison ML. Nivolumab for Recurrent Squamous-Cell Carcinoma of the Head and Neck. N Engl J Med. 2016 Nov 10;375(19):1856-1867. doi: 10.1056/NEJMoa1602252. Epub 2016 Oct 8. PMID 27718784
- [Background] Brahmer J, Reckamp KL, Baas P, Crino L, Eberhardt WE, Poddubskaya E, Antonia S, Pluzanski A, Vokes EE, Holgado E, Waterhouse D, Ready N, Gainor J, Aren Frontera O, Havel L, Steins M, Garassino MC, Aerts JG, Domine M, Paz-Ares L, Reck M, Baudelet C, Harbison CT, Lestini B, Spigel DR. Nivolumab versus Docetaxel in Advanced Squamous-Cell Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Jul 9;373(2):123-35. doi: 10.1056/NEJMoa1504627. Epub 2015 May 31. PMID 26028407
- [Background] Zhang J, Fang W, Qin T, Yang Y, Hong S, Liang W, Ma Y, Zhao H, Huang Y, Xue C, Huang P, Hu Z, Zhao Y, Zhang L. Co-expression of PD-1 and PD-L1 predicts poor outcome in nasopharyngeal carcinoma. Med Oncol. 2015 Mar;32(3):86. doi: 10.1007/s12032-015-0501-6. Epub 2015 Feb 22. PMID 25702326
- [Background] Lee VH, Lo AW, Leung CY, Shek WH, Kwong DL, Lam KO, Tong CC, Sze CK, Leung TW. Correlation of PD-L1 Expression of Tumor Cells with Survival Outcomes after Radical Intensity-Modulated Radiation Therapy for Non-Metastatic Nasopharyngeal Carcinoma. PLoS One. 2016 Jun 24;11(6):e0157969. doi: 10.1371/journal.pone.0157969. eCollection 2016. PMID 27341634
- [Background] Hsu C, Lee SH, Ejadi S, Even C, Cohen RB, Le Tourneau C, Mehnert JM, Algazi A, van Brummelen EMJ, Saraf S, Thanigaimani P, Cheng JD, Hansen AR. Safety and Antitumor Activity of Pembrolizumab in Patients With Programmed Death-Ligand 1-Positive Nasopharyngeal Carcinoma: Results of the KEYNOTE-028 Study. J Clin Oncol. 2017 Dec 20;35(36):4050-4056. doi: 10.1200/JCO.2017.73.3675. Epub 2017 Aug 24. PMID 28837405
- [Background] Ma BBY, Lim WT, Goh BC, Hui EP, Lo KW, Pettinger A, Foster NR, Riess JW, Agulnik M, Chang AYC, Chopra A, Kish JA, Chung CH, Adkins DR, Cullen KJ, Gitlitz BJ, Lim DW, To KF, Chan KCA, Lo YMD, King AD, Erlichman C, Yin J, Costello BA, Chan ATC. Antitumor Activity of Nivolumab in Recurrent and Metastatic Nasopharyngeal Carcinoma: An International, Multicenter Study of the Mayo Clinic Phase 2 Consortium (NCI-9742). J Clin Oncol. 2018 May 10;36(14):1412-1418. doi: 10.1200/JCO.2017.77.0388. Epub 2018 Mar 27. PMID 29584545
- [Background] Xiao WW, Huang SM, Han F, Wu SX, Lu LX, Lin CG, Deng XW, Lu TX, Cui NJ, Zhao C. Local control, survival, and late toxicities of locally advanced nasopharyngeal carcinoma treated by simultaneous modulated accelerated radiotherapy combined with cisplatin concurrent chemotherapy: long-term results of a phase 2 study. Cancer. 2011 May 1;117(9):1874-83. doi: 10.1002/cncr.25754. Epub 2010 Nov 16. PMID 21509764
- [Background] Lai SZ, Li WF, Chen L, Luo W, Chen YY, Liu LZ, Sun Y, Lin AH, Liu MZ, Ma J. How does intensity-modulated radiotherapy versus conventional two-dimensional radiotherapy influence the treatment results in nasopharyngeal carcinoma patients? Int J Radiat Oncol Biol Phys. 2011 Jul 1;80(3):661-8. doi: 10.1016/j.ijrobp.2010.03.024. Epub 2010 Jul 17. PMID 20643517
- [Background] Lee AW, Ng WT, Pan JJ, Poh SS, Ahn YC, AlHussain H, Corry J, Grau C, Gregoire V, Harrington KJ, Hu CS, Kwong DL, Langendijk JA, Le QT, Lee NY, Lin JC, Lu TX, Mendenhall WM, O'Sullivan B, Ozyar E, Peters LJ, Rosenthal DI, Soong YL, Tao Y, Yom SS, Wee JT. International guideline for the delineation of the clinical target volumes (CTV) for nasopharyngeal carcinoma. Radiother Oncol. 2018 Jan;126(1):25-36. doi: 10.1016/j.radonc.2017.10.032. Epub 2017 Nov 15. PMID 29153464
- [Background] Lee NY, Zhang Q, Pfister DG, Kim J, Garden AS, Mechalakos J, Hu K, Le QT, Colevas AD, Glisson BS, Chan AT, Ang KK. Addition of bevacizumab to standard chemoradiation for locoregionally advanced nasopharyngeal carcinoma (RTOG 0615): a phase 2 multi-institutional trial. Lancet Oncol. 2012 Feb;13(2):172-80. doi: 10.1016/S1470-2045(11)70303-5. Epub 2011 Dec 15. PMID 22178121
- [Background] Lee N, Harris J, Garden AS, Straube W, Glisson B, Xia P, Bosch W, Morrison WH, Quivey J, Thorstad W, Jones C, Ang KK. Intensity-modulated radiation therapy with or without chemotherapy for nasopharyngeal carcinoma: radiation therapy oncology group phase II trial 0225. J Clin Oncol. 2009 Aug 1;27(22):3684-90. doi: 10.1200/JCO.2008.19.9109. Epub 2009 Jun 29. PMID 19564532
- [Result] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Result] Keir ME, Butte MJ, Freeman GJ, Sharpe AH. PD-1 and its ligands in tolerance and immunity. Annu Rev Immunol. 2008;26:677-704. doi: 10.1146/annurev.immunol.26.021607.090331. PMID 18173375
- [Result] Latchman Y, Wood CR, Chernova T, Chaudhary D, Borde M, Chernova I, Iwai Y, Long AJ, Brown JA, Nunes R, Greenfield EA, Bourque K, Boussiotis VA, Carter LL, Carreno BM, Malenkovich N, Nishimura H, Okazaki T, Honjo T, Sharpe AH, Freeman GJ. PD-L2 is a second ligand for PD-1 and inhibits T cell activation. Nat Immunol. 2001 Mar;2(3):261-8. doi: 10.1038/85330. PMID 11224527
- [Result] Barber DL, Wherry EJ, Masopust D, Zhu B, Allison JP, Sharpe AH, Freeman GJ, Ahmed R. Restoring function in exhausted CD8 T cells during chronic viral infection. Nature. 2006 Feb 9;439(7077):682-7. doi: 10.1038/nature04444. Epub 2005 Dec 28. PMID 16382236